CLINICAL TRIAL: NCT07156162
Title: Comparing the Effectiveness of Taste vs. Health-Based Messaging Using Nutrition Education Videos on Increasing Herb and Spice Use to Improve Diet Quality
Brief Title: Effectiveness of Taste vs. Health-Based Messaging to Improve Diet Quality
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Travis Masterson, Assistant Professor, Penn State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: STUDY00027796
Record Dates: First submitted 2025-09-03; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Behavior, Health
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Taste video viewing participants followed by health video viewing participants (n=200) (Active Comparator): Participants in this arm will first watch the taste messaging focused videos, followed by the health messaging focused videos.
  Interventions: Other: Videos: Taste vs Health
- Health video viewing participants followed by taste video viewing participants (n=200) (Active Comparator): Participants in this arm will first watch the health messaging focused videos, followed by the taste messaging focused videos.
  Interventions: Other: Health vs. Taste

INTERVENTIONS:
Other: Videos: Taste vs Health — Participants in this intervention will watch taste and health focused messaging videos to determine which version is better suited to improve herb and spice usage to improve diet quality in American adults.
  Arms: Taste video viewing participants followed by health video viewing participants (n=200)
Other: Health vs. Taste — Participants in this intervention will watch health and taste focused messaging videos to determine which version is better suited to improve herb and spice usage to improve diet quality in American adults.
  Arms: Health video viewing participants followed by taste video viewing participants (n=200)

SUMMARY:
The purpose of this study is to compare the effectiveness of taste vs. health messaging using nutrition education videos. The investigators aim to compare and test 2 taste-based messaging vs. 2 health-based messaging that translate previous findings of how spices can improve diet quality. These objectives will be pursued via the following hypothesis:

Hypothesis 1: Are taste messaging videos more effective in improving consumer interest, knowledge, and confidence in using herbs and spices compared to health messaging focused videos? Hypothesis 2: Will consumers rate the taste messaging videos higher for liking, engagement, and acceptability of herbs and spices compared to health messaging focused videos?

DETAILED DESCRIPTION:
Participants will be randomly assigned to one of two groups: the first group (n~200) will view two taste messaging focused videos emphasizing taste and flavor first followed by the two health messaging focused videos. The second group (n~200) will receive the two health messaging focused videos emphasizing the importance of using herbs to improve health first followed by the two taste messaging focused videos. Randomization will occur using R and the randomization feature will be embedded in the survey. Both groups will have access to the same educational content but the time of viewing the messaging video will differ according to the taste or health focused arm. Participants will complete screening questions first, and if eligible, an online consent form. Participants will also complete an evaluation questionnaire after watching the taste messaging focused videos and after watching the health messaging focused videos. After participants have completed those questionnaires, they will be provided with a list of measures on why they liked a video and will be able to select if they preferred one over the other, as well as their feedback on the videos, and a demographics questionnaire. Investigators will use participants responses for analysis. All participants will complete the survey questions online using their own device.

ELIGIBILITY:
Inclusion Criteria:

* Adults, 18-75 years of age
* Reside in the United States
* Fluent in English
* Able to cook at home at least 2x/week or more

Exclusion Criteria:

* Outside of the 18-75 year age range
* Resides outside the United States
* Are not fluent in English
* Unable to cook at home at least 2x/week

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
1. Evaluation questionnaire for the taste videos and the health videos using a visual analog scale from "strongly disagree" to "strongly agree". | Right after watching the second set of nutrition education videos.

CONTACTS AND LOCATIONS:
Locations (1):
- Dynata Online Market Research Agency, Shelton, Connecticut, United States